CLINICAL TRIAL: NCT01349725
Title: A Safety Study of ARRY-502 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Array Biopharma, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Array BioPharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ARRAY-502-102
Record Dates: First submitted 2011-05-05; First posted 2011-05-09 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Healthy
Keywords: Safety

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARRY-502 (Experimental)
  Interventions: Drug: ARRY-502
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARRY-502 — Oral; multiple dose, escalating
  Arms: ARRY-502
Drug: Placebo — Oral; matching placebo
  Arms: Placebo

SUMMARY:
This is a Phase 1 study, involving a 14-day dosing period, designed to test the safety of investigational study drug ARRY-502 in healthy subjects. Approximately 32 healthy subjects from the United States will be enrolled in this study.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy male or female between the ages of 18 and 50 years.
* Females must be of nonchildbearing potential.
* Body mass index (BMI) of 18 to 32 and a total body weight > 50 kg (110 lbs) and < 114 kg (250 lbs).
* Additional criteria exist.

Key Exclusion Criteria:

* Evidence or history of clinically significant disease (excepting allergic rhinitis).
* Evidence of hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
* Gastrointestinal surgery that may interfere with motility or absorption.
* Serious illness requiring hospitalization within the previous 6 months.
* A positive test for drugs or alcohol.
* Recent use of tobacco- or nicotine-containing products. Use of any medications, grapefruit or supplements within the previous 14 days.
* Use of corticosteroids within the previous 28 days.
* Recent history of blood, plasma or platelet donation.
* Treatment with a small-molecule investigational drug within the previous 30 days or any biologic therapy within the previous 6 months.
* Prior exposure to investigational study drug ARRY-502.
* Additional criteria exist.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Characterize the safety profile of the study drug as determined by adverse events, clinical laboratory tests, electrocardiograms and vital signs. | 3 weeks
Characterize the pharmacokinetics of the study drug and metabolite as determined by plasma concentrations. | 2 weeks

SECONDARY OUTCOMES:
Characterize the pharmacodynamics of the study drug as determined by laboratory assays. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Madison, Wisconsin, United States